CLINICAL TRIAL: NCT06059287
Title: The Effect of Henagliflozin and Metformin on Myocardial Tissue-level Characteristics in Patients With Type 2 Diabetes and Obesity: A Prospective, Randomized, Open-label, Active Drug Controlled Clinical Trial
Brief Title: The Effect of Henagliflozin and Metformin on Myocardial Tissue-level Characteristics
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Jing Ma, Executive Officer of Endocrinology Department, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2023-0180
Record Dates: First submitted 2023-09-21; First posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Obesity; Type 2 Diabetes; Sodium-glucose Co-transporter-2 Inhibitor; Myocardial Fibrosis; Magnetic Resonance Imaging
Keywords: Metformin
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2 | interventions — henagliflozin; Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Henagliflozin (Experimental): Henagliflozin 10mg qd po
  Interventions: Drug: Henagliflozin
- Metformin (Active Comparator): Metformin 1000mg bid po
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Henagliflozin — Henagliflozin 10mg qd po
  Other Names: SHR3824
  Arms: Henagliflozin
Drug: Metformin — Metformin 1000mg bid po
  Other Names: Metformin Hydrochloride
  Arms: Metformin

SUMMARY:
This is a prospective, randomized, open-label, active drug controlled clinical trial that aims to compare the effects of henagliflozin or metformin on myocardial tissue level characteristics in type 2 diabetes patients with obesity. Eligible subjects with type 2 diabetes before randomisation and fulfilling all of the inclusion criteria and none of the exclusion criteria will be randomised in a 1:1 ratio to henagliflozin 10 mg once a day or metformin 1000 mg twice a day and treated for 24 weeks. The study includes five visits.

DETAILED DESCRIPTION:
MRI scanning will be assessed at baseline and at the end of the treatment period in order to to assess the cardiac morphology, cardiac function, and myocardial tissue characteristics. The cardiac MRI examination will be performed in accordance with a pre-defined MRI protocol. Images from all sites will be analyzed centrally at the core-lab using a dedicated software package and certified analysts.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with type 2 diabetes newly diagnosed based on the WHO (1999) criteria;
* Hemoglobin A1c levels >=7.0% and <=8.0%;
* Females or males ≥18 years up to 75 years of age.

Exclusion Criteria:

* Females or males <18 years.
* Clinical diagnosis of type 1 diabetes and other types of diabetes.
* Blood pressure at screening that would require a change in blood pressure treatment over the study period.
* History of stroke or other clinically significant cerebrovascular disease.
* Any of the following cardiovascular diseases:

  1. Atrial fibrillation, or other unstable or severe arrhythmia affecting heart function
  2. Unstable heart failure or any heart failure with NYHA class III and IV
  3. Significant valvular disease
  4. Significant peripheral artery disease
* Active malignancy requiring treatment at the time of visit 0.
* Patients with severe hepatic impairment.
* Unstable or rapidly progressing renal disease.
* Ongoing treatment with loop diuretics.
* Estimated Glomerular Filtration Rate (eGFR) <45 mL/min/1.73 m2.
* Women who has a positive pregnancy test at enrolment or randomization, or are breastfeeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Extra-cellular volume fraction | baseline and week 24
  To compare the effects of henagliflozin and metformin on extra-cellular volume fraction

SECONDARY OUTCOMES:
Mean Change in HbA1c Levels | baseline and week 24
  To compare the effects of henagliflozin and metformin on HbA1c Levels
Mean change in body mass index | baseline and week 24
  To compare the effects of henagliflozin and metformin on body mass index
Mean change in blood pressure | baseline and week 24
  To compare the effects of henagliflozin and metformin on blood pressure
Mean change in level of Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | baseline and week 24
  To compare the effects of henagliflozin and metformin on level of Homeostatic Model Assessment of Insulin Resistance
Native T2 mapping | baseline and week 24
  To compare the effects of henagliflozin and metformin on native T2 mapping

CONTACTS AND LOCATIONS:
Overall Officials: Jing Ma, Principal Investigator — RenJi Hospital

IPD SHARING:
Plan to Share IPD: No